CLINICAL TRIAL: NCT04149678
Title: A Phase 1, Randomized, Parallel-group, Open-label Study to Evaluate the Effect of Cyclosporine on the Single-dose Pharmacokinetics of Ozanimod and Major Active Metabolites in Healthy Adult Subjects
Brief Title: Drug Interaction Study of the Effect on Cyclosporine on Ozanimod and Major Active Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPC-1063-CP-001; U1111-1239-1156 (Other: WHO)
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Subjects; Ozanimod; Cyclosporine
MeSH Terms: interventions — ozanimod; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A - Ozanimod (Experimental): Subjects will receive a single oral dose of ozanimod 0.46 mg
  Interventions: Drug: Ozanimod
- Treatment Group B - Ozanimod plus Cyclosporine (Experimental): Subjects will receive a single oral dose of ozanimod 0.46 mg plus a single oral dose of cyclosporine 600 mg
  Interventions: Drug: Ozanimod; Drug: Cyclosporine

INTERVENTIONS:
Drug: Ozanimod — Ozanimod
Drug: Cyclosporine — Cyclosporine
  Arms: Treatment Group B - Ozanimod plus Cyclosporine

SUMMARY:
This is a Phase 1, randomized, parallel-group, open-label study. Forty subjects will be enrolled and will be randomized into 1 of the 2 treatment groups, with 20 subjects in each treatment group(sex will be used as a stratifying factor) as follows:

* Treatment Group A (reference): A single oral dose of ozanimod 0.46 mg
* Treatment Group B (test): A single oral dose of ozanimod 0.46 mg plus a single oral dose of cyclosporine 600 mg

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is a man or non-pregnant, non-lactating woman, ≥ 18 and ≤ 55 years of age at the time of signing the informed consent form (ICF).
2. Female subjects must meet at least 1 of the following criteria:

   * Negative serum pregnancy test at Screening and Day -1 (females of child-bearing potential [FCBP] only).
   * Postmenopausal (defined as 2 years after the last period and follicle-stimulating hormone [FSH] > 40 IU/L).
   * Received surgical sterilization (eg, bilateral tubal ligation, bilateral oophorectomy, hysterectomy) at least 6 months before Screening with medical records.
3. Female subjects of child-bearing potential must agree to practice a highly effective method of contraception throughout the study until completion of the follow-up phone call. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly. Acceptable methods of birth control in this study are the following:

   * Combined hormonal (oestrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.
4. Subject has a body weight of at least 110 pounds (50 kg); body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive (Screening and Day -1).
5. Subject is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, physical examination, clinical laboratory tests, and vital signs.
6. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
7. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject with a seated blood pressure outside 90 to 140 mmHg systolic or 50 to 90 mmHg diastolic at Screening or Day -1.
2. Subject with a seated pulse rate outside 55 to 90 beats per minute (bpm) at Screening or Day -1.
3. Subject has a presence or history of any abnormality or illness that, in the opinion of the investigator, may affect absorption, distribution, metabolism, or elimination of the IP (or would limit the subject's ability to participate in and complete this clinical study.
4. Subject has any condition that confounds the ability to interpret data from the study.
5. Subject has a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
6. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
7. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, vape, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) or marijuana (cigarette, joint, vape, edibles, etc) within 3 months prior to the first dose of IP.
8. Subject has a positive urine drug test including cotinine at Screening or Day -1.
9. Subject has a positive alcohol urine or breath test at Screening or Day -1.
10. Subject has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
11. Subject has used any systemic over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement (excluding vitamins/multivitamins) within 7 days prior to the first dose of IP. Herbal supplements including St. John's wort must be discontinued at least 28 days prior to the first dose of IP.
12. Subject has consumed pomelo-variety citrus fruits or juice (including pomelo, grapefruit, Seville oranges) within 7 days prior to the first dose of IP.
13. Subject has used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to the first dose of IP.
14. Subject has ingested alcohol within 7 days prior to the first dose of IP.
15. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to the first dose of IP.
16. Subject has poor peripheral venous access.
17. Subject has donated greater than 400 mL of blood within 60 days prior to Day 1.
18. Subject has history of hypersensitivity or allergic reaction to sphingosine 1-phosphate (S1P) receptor modulators or cyclosporine.
19. Subject with history of any medical condition or medical history that, in the opinion of the investigator, might confound the results of the study or jeopardize the safety or welfare of the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax | Up to approximately 15 days
  Maximum observed plasma concentration
Pharmacokinetic - AUC∞ | Up to approximately 15 days
  Area under the concentration-time curve from time 0 to infinity
Pharmacokinetic - AUClast | Up to approximately 15 days
  Area under the concentration-time curve from time 0 to time of last quantifiable concentration

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until 60 days after ozanimod dosing
  Number of participants with adverse event
Pharmacokinetic - Tmax | Up to approximately 15 days
  Time to Cmax
Pharmacokinetic - CL/F | Up to approximately 15 days
  Apparent oral clearance
Pharmacokinetic - Vz/F | Up to approximately 15 days
  Apparent volume of distribution during terminal phase after oral administration
Pharmacokinetic - t1/2 | Up to approximately 15 days
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/